CLINICAL TRIAL: NCT03443336
Title: Prospective Multi-center Surveillance Study on the Prevalence of Azole-resistant Aspergillus Spp. in Clinical Isolates ot Patients With Pulmonary Colonization or Invasive Infections in Switzerland
Brief Title: Azole-resistance in Aspergillus
Status: Completed | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Other Study IDs: 2017-00984; me17Khanna
Record Dates: First submitted 2018-02-09; First posted 2018-02-23 (Actual); Last update posted 2021-06-03 (Actual); Status verified 2021-06

CONDITIONS: Pulmonary Aspergillosis
MeSH Terms: conditions — Pulmonary Aspergillosis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — clinical Aspergillus spp. isolates
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Prospective multi-center surveillance study on the prevalence of azole-resistant Aspergillus spp. in clinical isolates of patients with pulmonary colonization or invasive infections in Switzerland

DETAILED DESCRIPTION:
Azole-resistance in Aspergillus (A.) fumigatus has emerged as a global health problem. Even more, it has been associated with high mortality rates in patients with invasive aspergillosis.

Generally, two routes of resistance development are distinguished either in patients with chronic pulmonary aspergillosis under long-term azole therapy or in agriculture by the use of azoles as fungicides.

The primary mechanisms of resistance that have been described in clinical strains include different point mutations in the cyp51A gene, which encodes the enzyme responsible for converting lanosterol to ergosterol via demethylation. Some resistant isolates also contain a tandem repeat in the promoter region of this gene that causes increased expression. These mutations, including TR34/L98H and TR46/Y121F/T289A have been identified in the environment and have been demonstrated to cause resistance to azole fungicides used in agriculture. These mutations were also recently identified in haematological patients suffering from invasive aspergillosis and were associated with a mortality rate of 88%.

Studies on the frequency of azole resistance in Aspergillus culture collections report the first resistant isolates up to 20 years earlier than clinical and environmental studies. Since then, microbiological resistance to azoles and clinical failures associated with this resistance have been reported in several countries in Europe and elsewhere. The United Kingdom and the Netherlands have reported increases in azole-resistant A. fumigatus. In the United Kingdom, a statistically significant increase in azole resistance was noted between 2004 and 2009, with rates of 5 to 7% in 2004 to 2006 increasing to up to 20% in 2009. These isolates were collected primarily in patients who received long-term azole therapy for the treatment of chronic pulmonary aspergillosis. The observation has increased the awareness of azole resistance in this patient population. Surveillance studies and case series over the last years suggest the global presence of azole resistance in A. fumigatus, including in Europe, the Middle East, Asia, Africa, Australia and, most recently, North and South America.

Moreover, some cryptic species of Aspergillus section Fumigati (e.g. A. lentulus, A. udagawae), which cannot be reliably distinguished from A. fumigatus by standard diagnostic methods, account for 3-5% of all A. fumigatus sensu lato clinical isolates and exhibit some level of intrinsic azole resistance. The proportion of these cryptic species in other Aspergillus sections (e.g. Flavi, Nigri, Terrei) is relatively unexplored. In addition, some rare Aspergillus species with intrinsic azole resistance, such as Aspergillus calidoustus (section Usti) are emerging as opportunistic pathogens in patients receiving azole prophylaxis. These cryptic or rare Aspergillus spp. are often misidentified because of the lack of discrimination by standard microbiological methods. Thus, their actual clinical relevance is unknown.

In Switzerland, comprehensive data on azole resistance in A. fumigatus are lacking. The major reason for this is the lack of routine testing of in vitro susceptibility of A. fumigatus isolates in most microbiology laboratories.

The Fungal Infections Network of Switzerland (FUNGINOS) offers an optimal platform to comprehensively assess the epidemiology of azole-resistance in A. fumigates and other Aspergillus spp. Only recently invasive Candida infections (candidemia) have been prospectively monitored by FUNGINOS over ten years from 2004 to 2013 in all Swiss University clinics and 20 University-affiliated hospitals.

ELIGIBILITY:
Inclusion Criteria:

* Available respiratory sample growing Aspergillus spp.
* Available clinical data

Exclusion Criteria:

• refusal to sign the general consent

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients with a respiratory sample growing Aspergillus spp., will be included
Sampling Method: Probability Sample
Enrollment: 400 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2021-06-02 (Actual)

PRIMARY OUTCOMES:
Azole-resistance in Aspergillus (A.) fumigatus | start of study until end of study (July 2017 until December 2018)
  Distribution of antifungal susceptibility profile of all tracheal and urinary samples in clinical Aspergillus isolates

CONTACTS AND LOCATIONS:
Overall Officials: Nina Khanna, Prof MD, Principal Investigator — University Hospital, Basel, Switzerland
Locations (1):
- Division of Infectious Diseases and Hospital Epidemiology, Basel, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided